CLINICAL TRIAL: NCT07326735
Title: MIRAGE Study: Clinical Outcomes of the Mamba Sirolimus-Eluting PTCA Balloon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frisch Medical Device Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRAGE-DCB-2023-01; MIRAGE-DCB-2023-01 (Other: Frisch Medical Devices Pvt Ltd)
Record Dates: First submitted 2025-12-10; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD))
Keywords: Drug Coated balloons, DCB , DEB, Sirolimus, de novo , in-stent restenosis lesions
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction; Color Vision Defects

STUDY DESIGN:
Intervention Model Description: Drug coted coronary PTCA balloons
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mamba Sirolimus Drug-Coated Balloon (DCB) (Experimental): Participants undergo percutaneous coronary angioplasty using the Mamba Sirolimus Drug-Coated Balloon (DCB) following standard lesion preparation. Balloon is inflated 30-45 seconds; multiple inflations permitted. No implant is left behind.
  Interventions: Device: Mamba Sirolimus-Eluting PTCA Balloon; Device: Percutaneous Coronary Angioplasty with Sirolimus-Coated Balloon

INTERVENTIONS:
Device: Mamba Sirolimus-Eluting PTCA Balloon — PTCA coronary angioplasty with Drug coated balloon for De novo and in stent restenosis cases
Device: Percutaneous Coronary Angioplasty with Sirolimus-Coated Balloon — Percutaneous transluminal coronary angioplasty performed using a sirolimus-coated balloon catheter intended to deliver the drug to the arterial wall during balloon inflation. The balloon is positioned across the target lesion following standard lesion preparation and inflated for approximately 30-45 seconds; multiple inflations are permitted. No permanent implant or scaffold remains in the artery. The sirolimus coating is designed to inhibit neointimal hyperplasia and support vessel healing, offering a "leave-nothing-behind" approach to treatment of obstructive coronary artery disease.

SUMMARY:
This Clinical Evaluation Report (CER) covers the Mamba Sirolimus-Eluting PTCA Balloon catheter intended for the treatment of coronary artery disease in de novo or in-stent restenosis lesions. It includes analysis of clinical data from the MIRAGE clinical study, literature data on sirolimus DCBs, bench and preclinical testing, and risk-benefit evaluation in compliance with MDR Annex XIV.

DETAILED DESCRIPTION:
This Clinical Evaluation Report (CER) covers the Mamba Sirolimus-Eluting PTCA Balloon catheter intended for the treatment of coronary artery disease in de novo or in-stent restenosis lesions. It includes analysis of clinical data from the MIRAGE clinical study, literature data on sirolimus DCBs, bench and preclinical testing, and risk-benefit evaluation in compliance with MDR Annex XIV.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Patient diagnosed with obstructive coronary artery disease suitable for percutaneous coronary intervention.
3. Target lesion located in a native coronary artery with reference vessel diameter of ≥2.0 mm.
4. Successful lesion preparation prior to DCB treatment (defined by <30% residual stenosis and TIMI flow ≥2).
5. Patient able and willing to comply with scheduled follow-up evaluations at 1, 6, and 12 months.
6. Signed informed consent obtained prior to the procedure.

Exclusion Criteria:

1. ST-elevation myocardial infarction (STEMI) within the previous 48 hours.
2. Left main disease >50% requiring stenting or surgical intervention.
3. Presence of thrombus or severe vessel calcification that prevents adequate balloon expansion.
4. Previous stenting at the target lesion within the previous 3 months.
5. Known allergy or contraindication to sirolimus, contrast media, or dual antiplatelet therapy.
6. Pregnant or breastfeeding women.
7. Life expectan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Composite Measure of Major Adverse Cardiac Events (MACE) at 12 Months including Cardiac Death, Myocardial Infarction, and Clinically Driven Target Lesion Revascularization | 12 Months
  MACE is defined as the composite rate of cardiac death, myocardial infarction, or clinically driven target lesion revascularization occurring within 12 months following the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavin Oza, Study Chair — Frisch Medical Devices
Locations (2):
- Prime Heart Institute, Yangon, Gujarat, Burma
- National Heart Centre Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT07326735/Prot_000.pdf